CLINICAL TRIAL: NCT04976777
Title: Evaluation of an Updated Dexamethasone Posterior Segment Drug Delivery System Applicator in Participants With Macular Edema Due to Retinal Diseases
Brief Title: A Study to Evaluate an Updated Dexamethasone Intravitreal (Into the Eye) Applicator in Adult Participants With Macular Edema Due to Diseases of the Retina
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1491-801-007
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Macular Edema
Keywords: Macular Edema; Dexamethasone; Branch Retinal Vein Occlusion; Central Retinal Vein Occlusion; Diabetic Macular Edema; Noninfectious Uveitis; Ozurdex; Dexamethasone Posterior Segment Drug Delivery System (DEX PS DDS)
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Updated Dexamethasone Posterior Segment Drug Delivery System (DEX PS DDS) 0.7 mg (Experimental): DEX PS DDS 0.7 mg implant was administered intravitreally into the study eye using updated applicator at Day 1 and followed until Day 7.
  Interventions: Device: Updated DEX PS DDS Applicator; Drug: Dexamethasone
- Approved DEX PS DDS 0.7 mg (Active Comparator): DEX PS DDS 0.7 mg implant was administered into the study eye using currently approved applicator at Day 1 and followed until Day 7.
  Interventions: Device: Approved DEX PS DDS Applicator; Drug: Dexamethasone

INTERVENTIONS:
Device: Updated DEX PS DDS Applicator — Intravitreal Administration
  Arms: Updated Dexamethasone Posterior Segment Drug Delivery System (DEX PS DDS) 0.7 mg
Device: Approved DEX PS DDS Applicator — Intravitreal administration
  Other Names: OZURDEX®
  Arms: Approved DEX PS DDS 0.7 mg
Drug: Dexamethasone — Dexamethasone 0.7 mg in a solid polymer drug delivery system

SUMMARY:
The Dexamethasone Posterior Segment Drug Delivery System (DEX PS DDS) Applicator is used to deliver an implant with medicine to the eye. AbbVie is updating the DEX PS DDS Applicator. This purpose of this study is to show that the updated DEX PS DDS Applicator works in adult participants with macular edema due to retinal diseases.

The DEX PS DDS is approved for the treatment of macular edema. Participants will be placed into 1 of 2 groups, called treatment arms. Each group receives the same treatment drug delivered using different applicators. Around 54 adult participants with macular edema will be enrolled in the study in approximately 7-10 sites in the United States.

Participants will receive a single intravitreal (into the eye) administration of DEX PS DDS implant using either the currently-approved DEX PS DDS Applicator or the the updated Applicator. The participants will be observed for a duration of 7 days, with the DEX PS DDS implant received on day 1 and follow-up through day 7.

The updates being evaluated in this study are related to the DEX PS DDS Applicator only, with the safety and efficacy of the DEX PS DDS implant well characterized and the same as the currently marketed product. Participants will attend regular visits during the study at a hospital or clinic. The applicator function will be checked by medical assessment, checking for side effects, procedural complications and/or product complaints, and evaluating the administration procedure.

ELIGIBILITY:
Inclusion Criteria:

- Participants with macular edema due to retinal vein occlusion (branch retinal vein occlusion or central retinal vein occlusion) or diabetic macular edema.

Exclusion Criteria:

- Participants with ocular conditions in the study eye for which Dexamethasone Posterior Segment Drug Delivery System Implant is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (7):
- United States (7):
  - Global Research Management /ID# 238944, Glendale, California
  - Advanced Eye Centers Inc /ID# 233429, North Dartmouth, Massachusetts
  - Discover Vision Centers /ID# 239366, Independence, Missouri
  - Charleston Neurosciences Institute /ID# 238521, Charleston, South Carolina
  - Retina Research Institute of Texas /ID# 231420, Abilene, Texas
  - Texas Retina Associates /ID# 231305, Arlington, Texas
  - North Texas Retina Consultants /ID# 241013, Willow Park, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 7 investigational sites in the United States from 12 October 2021 to 7 February 2022.
Period: Overall Study
Arm/Group | Updated Dexamethasone Posterior Segment Drug Delivery System (DEX PS DDS) 0.7 mg | Approved DEX PS DDS 0.7 mg
Started | 36 | 18
Completed | 35 | 18
Not Completed | 1 | 0
Not completed — COVID-19 Infection | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included of all participants who received DEX PS DDS Implant.
Groups:
- Updated DEX PS DDS 0.7 mg: DEX PS DDS 0.7 mg implant was administered intravitreally into the study eye using updated applicator at Day 1 and followed until Day 7.
- Total: Total of all reporting groups
Arm/Group | Updated DEX PS DDS 0.7 mg | Approved DEX PS DDS 0.7 mg | Total
Number analyzed (Participants) | 36 | 18 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (11.04) | 65.3 (11.94) | 65.9 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 20 | 7 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 29 | 15 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 33 | 16 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing at Least One Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.
Time Frame: Up to 7 Days After Study Drug Administration
Population: SAS included of all participants who received DEX PS DDS Implant.
Measure: Count of Participants; unit: Participants
Arm/Group | Updated DEX PS DDS 0.7 mg | Approved DEX PS DDS 0.7 mg
Number analyzed (Participants) | 36 | 18
Participants | 13 | 7

2. Other Pre Specified Outcome: Dexamethasone Posterior Segment Drug Delivery System (DEX PS DDS) Updated Applicator Performance
Description: The investigator evaluated whether the updated DEX PS DDS Applicator dispensed the DEX PS DDS implant in the vitreous cavity and performed as intended, using a treatment administration assessment form.
Time Frame: Day 1 After Study Drug Administration
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 7 Days After Study Drug Administration
Arm/Group | Updated DEX PS DDS 0.7 mg | Approved DEX PS DDS 0.7 mg
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/18
Other Adverse Events (participants affected / at risk) | 11/36 | 7/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Updated DEX PS DDS 0.7 mg (N=36) | Approved DEX PS DDS 0.7 mg (N=18)
COVID-19 PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Updated DEX PS DDS 0.7 mg (N=36) | Approved DEX PS DDS 0.7 mg (N=18)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 10 (10) | 7 (7)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT04976777/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT04976777/SAP_001.pdf